CLINICAL TRIAL: NCT00822198
Title: The Effect of Plantar Vibration on the Progression of Peripheral Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Binghamton University (Other)
Collaborators: NY State Office of Science, Technology and Academic Research (NYSTAR) (Unknown)
Responsible Party: Leann Lesperance, Binghamton University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 240-05
Record Dates: First submitted 2009-01-13; First posted 2009-01-14 (Estimated); Last update posted 2009-01-14 (Estimated); Status verified 2009-01

CONDITIONS: Peripheral Neuropathy
Keywords: peripheral neuropathy; diabetes; plantar vibration
MeSH Terms: conditions — Peripheral Nervous System Diseases; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- plantar vibration (Experimental): Subject will use Juvent plantar vibration device daily in the home or office for six months.
  Interventions: Device: plantar vibration

INTERVENTIONS:
Device: plantar vibration — Subjects in the experimental component of the trial will be provided with a Juvent 1000-CS device in their home or workplace. The device will be placed in a convenient location where the device does not represent a trip hazard, and yet is readily accessible for use. The subjects will be instructed to use the device whenever it is convenient to do so, either by standing on the device, or by sitting with their feet on the device. Downloads of usage data will be obtained intermittently. Period interviews with the subjects will be conducted to ensure that the device is operating and that no problems are encountered with device usage.

SUMMARY:
The purpose of this study is to assess the effect of vibration of the plantar surface of the foot on peripheral neuropathy.

DETAILED DESCRIPTION:
Background: Peripheral neuropathy has a prevalence approaching 10% in the general population. The pathophysiology of peripheral neuropathy is poorly understood or undetermined. While many causes of peripheral neuropathy are known, a significant number of cases are idiopathic. The most common cause of neuropathy relates to glucose intolerance or overt diabetes. Exogenous factors such as smoking constrict small cutaneous blood vessels, thereby inhibiting small nerve fiber nutrition. Symptoms of neuropathy include numbness, pain, difficulty with balance, lack of temperature perception, and weakness which can lead to significant disability. Classification of neuropathies can be made based on nerve fiber size: large fiber, small fiber and mixed large and small fiber types. Plantar vibration which affects large fibers has been demonstrated to enhance peripheral and systemic blood flow, peripheral lymphatic and venous drainage (Stewart, Karman, Montgomery, & McLeod, 2005). Since fluid retention in axons, nerve sheaths and surrounding connective tissues may contribute to neuropathy, it is hypothesized that plantar vibration may repair the small peripheral fibers, thereby improving the symptoms of neuropathy.

Purposes:

1. To assess the effect of plantar vibration on regeneration of small peripheral nerve fibers, peripheral neuropathy and quality of life in patients with diagnosed peripheral neuropathy.
2. To assess the correlation of health history, demographic variables, diet, alcohol and smoking history with small fiber neuropathy analysis by skin biopsy and plantar vibration.

Design: The study will employ a cross-over experimental design with subjects acting as their own controls. Independent variables are the plantar stimulation (intervention), and the characteristics of the subjects that include health history, demographic variables, self reported diet, alcohol, and smoking history, as well as urinary cotinine (a quantitative measure of smoking history). The dependent variables are the assay of intraepidermal nerve fibers in small-fiber neuropathy, clinical assessment of peripheral neuropathy, serum levels of Hgb A1C, and quality of life measurement.

ELIGIBILITY:
Inclusion Criteria:

* Clinical evidence of neuropathy
* Normal to moderate evidence of neuropathy on nerve conduction studies

Exclusion Criteria:

* Currently on medications with a known risk of neuropathy
* Pregnant
* Evidence of peripheral vascular disease

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-03; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
intraepidermal nerve fiber density in ankle and thigh | 0, 6 and 12 months

SECONDARY OUTCOMES:
quality of life score | 0, 6 and 12 months
clinical assessment of peripheral neuropathy | 0, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Leann M Lesperance, MD, PhD, Principal Investigator — Binghamton University
Locations (1):
- Neurology Associates, Corning, New York, United States